CLINICAL TRIAL: NCT06295874
Title: Effect of Aromatherapy Massage Applıed to Intensıve Care Patıents on Physıologıcal Parameters, Paın, Anxıety and Intensıve Care Comfort
Brief Title: The Effect of Aromatherapy Massage on Pain, Anxiety and Comfort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nilgün Erdoğan (Other)
Responsible Party: Sponsor-Investigator, Nilgün Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Organization: Nigde Omer Halisdemir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12.10.2022/50
Record Dates: First submitted 2024-02-02; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; High Blood Pressure; Stroke, Ischemic
Keywords: intensive care; pain; anxiety; comfort; aromatherapy massage
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Hypertension; Ischemic Stroke; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled single blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): After obtaining written and verbal permission from the families of the patients in the intervention group by signing the Informed Volunteer Consent Form, the patients were filled out the Patient Introduction Form, Patient Monitoring Form and Medication Monitoring Form by the nurses. The massage process, which was performed according to the application protocol of the aroma oil prepared for the patients (5 drops of lavender oil, 4 drops of thyme oil, 3 drops of eucalyptus oil and 20 ml of almond oil in 20 ml), was performed by the researcher by stroking the patient's back and chest, effleurage, re-effleurage, back massage. Deep caressing and stroking on the dorsal surface were performed in 6 consecutive steps.
  Interventions: Other: Effect of aromatherapy massage on vital signs, pain, anxiety and comfort level
- Placebo Control Group (Placebo Comparator): After obtaining written and verbal approval from the families of the patients included in the placebo control group by signing the Informed Volunteer Consent Form, the patients were filled out the Patient Introduction Form, Patient Monitoring Form and Medication Monitoring Form by the nurses. According to the oil application protocol, the massage with almond oil was performed by the researcher in 6 consecutive steps by stroking the patient's back and chest, effleurage, re-effleurage, deep stroking of the back and stroking the back surface.
  Interventions: Other: Effect of aromatherapy massage on vital signs, pain, anxiety and comfort level

INTERVENTIONS:
Other: Effect of aromatherapy massage on vital signs, pain, anxiety and comfort level — The study applied a mixture of lavender, thyme and eucalyptus oil (5 drops of lavender oil, 4 drops of thyme oil, 3 drops of eucalyptus oil and 20 ml of almond oil in 20 ml) to patients who were monitored in intensive care on high-flow and oxygen, for three days. It was conducted as a randomized controlled single-blind study to evaluate the effects of aromatherapy massage applied twice a day for a total of 30 minutes on some physiological parameters, pain, anxiety and comfort levels.

SUMMARY:
Patients in the intensive care unit (ICU) experience physical and psychological discomfort, including pain. Anxiety is a condition frequently encountered in the ICU. The hospital environment, especially the ICU, is reported as a significant cause of anxiety for patients. Comfort is a holistic, subjective and multidimensional concept that is affected by physical, environmental, social and psycho-spiritual contexts and changes over time and space. Comfort in intensive care is often associated with pain relief and end-of-life care. Assessment tools have been developed to measure patient comfort in the ICU, including levels of pain, delirium, and sedation. This work; Patients who are monitored in intensive care under high-flow and oxygen are treated with a mixture of lavender, thyme and eucalyptus oil (20 ml; lavender oil 5 drops, thyme oil 4 drops, eucalyptus oil 3 drops and 20 ml almond oil) twice a day for three days. This study was conducted to determine the effect of aromatherapy massage applied for a total of 30 minutes on some physiological parameters, pain, anxiety and intensive care comfort of the patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over,
* Conscious patients,
* Staying in intensive care for 24 hours or more,
* Those with stable hemodynamic status,
* Receiving O2 therapy,
* Intubated patients, patients who have passed 24 hours after being extubated,
* Those whose saturation level is 85 and above

Exclusion Criteria:

* Patients with peripheral neuropathy or quadriplegia,
* Patients with open wounds on their body,
* Patients receiving analgesia and sedation infusion,
* Patients who are sedated,
* Patients in delirium,
* Patients with an allergy detected before starting the application,
* Patients with a GKS (Glasgow Coma Scale) score of 3 and below

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Patient Introduction Form | 2 years
  The "Patient Introduction Form" prepared by the researcher based on the literature in order to obtain information about the characteristics of the patients who will form the sample includes questions such as the medical diagnosis of the patients, age, gender, chronic diseases, length of stay in intensive care, use of analgesics and sedative drugs.

SECONDARY OUTCOMES:
Patient Follow-up Form | 2 years
  The patient follow-up form was created by the researcher, and the follow-up results of physiological parameters throughout the study will be included in the form. Vital signs and oxygen saturation results of the patients before and after the application will be recorded on the patient follow-up form by the nurses who collect the data of the study.

OTHER OUTCOMES:
Drug Monitoring Form | 2 years
  The medication monitoring form was created by the researcher, and the form will include the dosage of the analgesic and sedative medications the patient received in the intensive care unit during the study. The medication monitoring form will be recorded with the dosage taken before and after the application by the nurses who collect the data of the study.
Visual Pain Scale | 2 years
  The scale developed by Price et al. (1983) is a scale in which patients evaluate their pain between 1 and 10. VAS is a scale used to describe varying degrees of pain experienced by a patient. It is evaluated at varying degrees between "0", "no pain" and "10", "severe pain".
Face Anxiety Scale | 2 years
  The Facial Anxiety Scale was developed to determine the presence and level of patient anxiety based on facial expressions. The Facial Anxiety Scale, developed by McKinley and colleagues (2003), has been used in several studies for patients on invasive and non-invasive ventilation. Each item in the anxiety subscale is rated between 1 and 5 points, ranging from "not at all" to "extremely".
Comfort Rating Scale | 2 years
  Numerik Konfor Derecelendirme Ölçeği, Kolcaba (2003) tarafından geliştirilen (Kolcaba, 2003), 0'dan 10'a kadar değişen derecelerde kullanılan bir analog skaladır. Rahatlık 0-10 arasında derecelendirilmektedir; 0, "hiç konfor yok", 10 "en yüksek konforu" göstermektedir. Hastanın durumuna göre değerlendirilmesi yapılmaktadır

CONTACTS AND LOCATIONS:
Locations (1):
- Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)